CLINICAL TRIAL: NCT00906256
Title: A Clinical Pharmacology Study to Determine the Pharmacokinetic, Safety and Tolerability Profile of Oral Doses of AZD7295 in Healthy Subjects
Brief Title: Clinical Pharmacology Study of AZD7295 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arrow Therapeutics (Industry)
Responsible Party: Dr Joanne Collier, Pharmaceutical Profiles Ltd
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: HCV689-103
Record Dates: First submitted 2009-05-11; First posted 2009-05-21 (Estimated); Last update posted 2010-02-12 (Estimated); Status verified 2010-02

CONDITIONS: Healthy
Keywords: Hepatitis C; Pharmacokinetics; AZD7295; Healthy volunteers
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AZD7295 (Active Comparator): AZD7295
  Interventions: Drug: AZD7295
- Placebo capsule (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD7295 — Capsules 260mg, 455mg, 650mg (single doses), 650mg q12h, 650mg q8h.
  Arms: AZD7295
Drug: Placebo — Placebo
  Arms: Placebo capsule

SUMMARY:
The purpose of this study is to determine the pharmacokinetic profile of oral doses of AZD7295 capsules in healthy subjects, and also to assess the effects of food as well as safety and tolerability.

DETAILED DESCRIPTION:
OBJECTIVES: Primary

* To determine the pharmacokinetic profiles of oral doses of AZD7295 capsules administered to healthy subjects
* To study the effect of food on the pharmacokinetic profiles of oral doses of AZD7295 capsules in healthy subjects
* To assess the safety and tolerability profiles of oral daily doses of AZD7295 capsules in healthy subjects TYPE AND DESIGN: Part A A phase I, single-centre, double-blind, randomised, placebo-controlled, crossover, food effect study in healthy subjects

Part B A phase I, single-centre, double-blind, randomised, placebo-controlled, ascending dose study in healthy subjects

NUMBER OF SUBJECTS: 16 subjects will take part in a total of 4 treatment periods.

SUBJECT CHARACTERISTICS: Healthy males and females of non-child bearing potential aged 18 to 65 years.

Recruitment will not be balanced for gender or any other variable.

TREATMENT: Part A

Subjects will be randomised to receive AZD7295 or placebo (14 active; 2 placebo) in either the fed or fasted state according to the treatment allocation:

Treatment A: 260 mg (4 x 65 mg) AZD7295 capsules or placebo dosed in the fed state

Treatment B: 260 mg (4 x 65 mg) AZD7295 capsules or placebo dosed in the fasted state

Following dosing of the first two periods there will be a period of interim analysis, during which the pharmacokinetic data will be reviewed in order to determine whether the remaining treatments will be dosed either in the fed or fasted state.

Subjects from Part A will continue into Part B of the study.

Part B

Subjects will be allocated to two groups of n=8 (Group 1 and Group 2) and randomised to receive AZD7295 or placebo (6 active; 2 placebo). Subjects will receive two of the ascending dose treatments in the following order according to group allocation:

Group 1:

Treatment C: 455 mg (7 x 65 mg) AZD7295 or placebo dosed either in the fed or fasted state;

Group 2:

Treatment D: 650 mg (10 x 65 mg) AZD7295 or placebo dosed either in the fed or fasted state;

Group 1:

Treatment E: 650 mg (10 x 65 mg) AZD7295 or placebo, twice a day (q12h) dosed either in the fed or fasted state (total administered dose: 1300 mg);

Group 2:

Treatment F: 650 mg (10 x 65 mg) AZD7295 or placebo, three times a day (q8h) dosed either in the fed or fasted state (total administered dose: 1950 mg).

Safety data and limited PK data will be reviewed by the data review group prior to proceeding to the next dose level.

During the dose escalation phase a maximum of 4 subjects will be dosed per day.

MAIN OUTCOME MEASURES: The primary outcome will be to determine the pharmacokinetic profiles of AZD7295 when dosed in the fed and fasted state and to assess the safety and tolerability of higher daily doses of AZD7295.

GENERAL SCHEDULE: Screening is planned to start in April 2009, with the clinical phase due to be completed by the end of July 2009

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or healthy females of non-child bearing potential
2. Aged 18-65 years;
3. Body Mass Index (BMI) of 18-32kg/m2;
4. Normal electrocardiograms (ECGs) or with clinically insignificant abnormalities in the opinion of the Investigator;
5. Normal vital signs or with clinically insignificant abnormalities in the opinion of the Investigator;
6. Clinically normal physical findings and safety laboratory values at the time of the screening visit, as judged by the Investigator;
7. Must be willing and able to participate in the whole study and must provide written informed consent.

Exclusion Criteria:

1. Participation in a clinical research study involving investigational drugs or dosage forms within the previous 3 months;
2. Subjects who have previously been enrolled in this study;
3. A past or current disease, which as judged by the Investigator, could affect the subject's participation in or the outcome of the study. These diseases include, but are not limited to cardiovascular disease, malignancy, hepatic disease, renal disease, haematological disease, neurological disease, immunological disease and endocrine disease;
4. Subjects who have ever sought advice from or been referred to a GP or counsellor for abuse or misuse of alcohol, non medical drugs, medicinal drugs or other substance abuse e.g. solvents;
5. Subjects who admit to any current or previous use of Class A drugs such as opiates, cocaine, ecstasy, lysergic acid diethylamide (LSD) and intravenous amphetamines (Subjects who admit to occasional past use of cannabis will not be excluded as long as they have a negative drugs of abuse test and have been abstinent for at least 12 months;);
6. Positive drugs of abuse test result (Appendix 1, Section 20);
7. Regular alcohol consumption in males >21 units per week and females >14 units per week (1 Unit = ½ pint beer, a 25 mL shot of 40% spirit or a 125 mL glass of wine);
8. Smoking of more than 10 cigarettes per day and the inability to refrain from smoking during confinement;
9. Females of child bearing potential, as detailed in Section 9.4;
10. Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the PI (Appendix 1, Section 20);
11. History of adverse reaction or allergy to study drug or its excipients. If the subject suffers from hayfever they must not have or be expecting to have symptoms during the study period;
12. Subjects with known present or past medical history, or family history (as far as known by the subject) of any of the following cardiovascular findings:

    * 2nd degree AV-block (type II) or 3rd degree AV-block and/or other relevant arrhythmias
    * Prolonged QT-interval syndrome or other cardiac conduction disorder QTc > 450 ms
    * PR interval outside range of 120 - 220 ms
    * Evidence of clinically significant T wave abnormalities
13. Donation of blood within the previous three months;
14. Subjects will be excluded from the study if they are considered by the PI to be at risk of transmitting, thorough blood or other body fluids, the agents responsible for acquired immunodeficiency syndrome (AIDS) or other sexually transmitted disease or hepatitis;
15. Positive HBV, HCV or HIV results;
16. Excessive use of caffeine (more than five cups of coffee or equivalent per day);
17. Subjects receiving prohibited medication as described in Section 9.5;
18. Subjects with planned surgery, dental procedure or hospitalisation during the study;
19. Failure to satisfy the PI of fitness to participate for any other reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To determine the pharmacokinetic profiles of oral doses of AZD7295 capsules administered to healthy subjects. | PK samples at pre-dose, 0.5h, 1.0h, 1.5h, 2.0h, 2.5h, 3.0h, 4.0h, 6.0h, 12.0h and 24.0h post dose.
To study the effect of food on the pharmacokinetic profiles of oral doses of AZD7295 capsules in healthy subjects | 1st two treatment days of study
To assess the safety and tolerability profiles of oral doses of AZD7295 in healthy subjects. | at each dosing day

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaceutical Profiles Ltd, Nottingham, United Kingdom